CLINICAL TRIAL: NCT04968574
Title: A Phase 2, Multi-Center Study Evaluating the Safety and Efficacy of ENV-101 (Taladegib) in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Study Evaluating the Safety and Efficacy of ENV-101 in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endeavor Biomedicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENV-IPF-101
Record Dates: First submitted 2021-06-29; First posted 2021-07-20 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: hedgehog; smoothened; pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis | interventions — LY2940680

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ENV-101 (Experimental): taladegib, 200 mg tablet, once daily for 12 weeks
  Interventions: Drug: taladegib
- placebo (Placebo Comparator): placebo, tablet, once daily for 12 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: taladegib — hedgehog pathway inhibitor dosed once daily
  Arms: ENV-101
Drug: placebo — identical tablets to the experimental arm with no active ingredient
  Arms: placebo

SUMMARY:
This is a Phase 2, randomized, placebo controlled, multi-center study in subjects with mild to moderate IPF. Eligible subjects will be randomized to receive placebo or ENV-101 as a daily oral dose for 12 consecutive weeks of treatment. Following treatment, subjects will be observed for an additional 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* IPF diagnosis based upon American Thoracic Association, Japanese Respiratory Society, European Respiratory Society, Latin American Thoracic Association guidelines within the last 7 years. Diagnosis will be confirmed to be consistent with IPF by centrally read high resolution computed tomography (HRCT).
* Ability to successfully perform lung function tests.
* Subjects are willing to remain on study treatment for the duration of the study.
* Subjects have a full understanding of the informed consent.

Exclusion Criteria:

* Evidence of other known causes of interstitial lung disease (ILD) (e.g., domestic, and occupational environmental exposures, connective tissue disease [CTD], and drug toxicity), lung transplant expected within 12 months of screening or evidence of clinically significant lung disease other than IPF including but not limited to asthma, chronic obstructive pulmonary disease (COPD), uncontrolled pulmonary hypertension and emphysema where computed tomography (CT)-assessed extent of emphysema is greater than extent of fibrosis.
* History of malignancy, including carcinoma during the preceding 5 years. With the following exceptions:

  1. Prior history of in situ basal or squamous cell skin cancer that was successfully treated with curative therapies.
  2. Subjects with other malignancies if they have been continuously disease free for at least 5 years prior to study start.
  3. Subjects with prostate cancer that are managed by surveillance are also eligible.
* Current use of supplemental oxygen for any condition unless prior approval is received from the Sponsor.
* Smoking within 6 months of study start, current smoker, or unwillingness to refrain from smoking during the clinical trial duration.
* Presence of active infection at study start or confirmed active human immunodeficiency virus (HIV), Hepatitis B virus (HBV) or Hepatitis C virus (HCV).
* Occurrence of serious illness requiring hospitalization within 90 days prior to study start.
* Current or previous use (within 30 days prior to study start) of the following:

  1. N-acetylcysteine
  2. endothelin receptor antagonist
  3. riociguat
  4. prostacyclin or prostacyclin analogue
  5. Warfarin for IPF
  6. Cytotoxic agents (e.g., colchicine if used for IPF)
  7. Radiation to the lungs
  8. Pulmonary rehabilitation
  9. Investigational agent for IPF
  10. Immunosuppressive medications (e.g., methotrexate, azathioprine)
  11. Systemic or inhaled glucocorticosteroids
  12. Antifibrotic therapy (e.g., nintedanib, pirfenidone)
* Regular use of phosphodiesterase type-5 inhibitor, occasional use for erectile dysfunction will be allowed.
* Use of drugs that are known moderate or stronger CYP3A4 inhibitors or inducers within 12 days prior to study start.
* Males and females of reproductive potential who are sexually active and unwilling to use birth control for the duration of the study and for 3 months after their final dose.
* Females that are pregnant or nursing.
* Females and males that are unwilling to refrain from blood or blood product donation for the duration of the study and for 30 days after their final study dose.
* Males who are unwilling to refrain from sperm donation and females who are unwilling to refrain from egg donation for the duration of the study and for 3 months after their final study dose.
* Subjects with a history of a severe allergic reaction or anaphylactic reaction or known hypersensitivity to any component of ENV-101.
* Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study investigative site or the study Sponsor.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in frequency of adverse events (AEs) | Baseline to Week 18
  An AE is any untoward medical occurrence in a study subject administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment under investigation. Frequency of a given AE is determined by dividing the total number of that AE observed during the study by the total number of subjects in the study.
Change from baseline in severity of AEs | Baseline to Week 18
  Severity of AEs are categorized as mild, moderate or severe as described below:
  * Mild - Events require minimal or no treatment and do not interfere with the subject's daily activities.
  * Moderate - Events result in a low level of inconvenience or concern with the therapeutic measures. Moderate events may cause some interference with functioning.
  * Severe - Events interrupt a subject's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually potentially life-threatening or incapacitating.
Change from baseline in vital sign measurements - pulse | Baseline to Week 18
  Comparison of a subject's pulse rate at the beginning of the study to that subject's pulse rate at the completion of the study.
Change from baseline in vital sign measurements - blood pressure | Baseline to Week 18
  Comparison of a subject's blood pressure at the beginning of the study to that subject's blood pressure at the completion of the study.
Change from baseline in vital sign measurements - respiration rate | Baseline to Week 18
  Comparison of a subject's respiration rate (number of breaths taken per minute while at rest) at the beginning of the study to that subject's respiration rate at the completion of the study.
Change from baseline in vital sign measurements - temperature | Baseline to Week 18
  Comparison of a subject's body temperature at the beginning of the study to that subject's body temperature at the completion of the study.
Change from baseline in blood oxygen saturation level | Baseline to Week 18
  Comparison of a subject's blood oxygen saturation level (measured at rest using a pulse oximeter) at the beginning of the study to that subject's blood oxygen saturation level at the completion of the study.
Incidence of clinical laboratory abnormalities | Baseline to Week 18
  Assessment of the clinical laboratory measurements (chemistry, hematology, urinalysis parameters) that are above or below the laboratory normal ranges. Incidence of clinical laboratory abnormalities is determined by dividing the total number of clinical laboratory abnormalities by the total number of subjects in the study.
Severity of clinical laboratory abnormalities | Baseline to Week 18
  Assessment of the severity (defined as either clinically significant or not clinically significant) for the clinical laboratory abnormalities observed during the study.
Number of hospitalizations | Baseline to Week 18
  Assessment of the number of hospitalizations for any reason observed among all subjects from the beginning of the study to the completion of the study.

SECONDARY OUTCOMES:
Change from baseline of FVC (forced vital capacity) | Baseline and Week 12
  FVC is the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible, as measured during a spirometry test.
Change from baseline of DLCO (diffusing capacity of the lungs for carbon monoxide) | Baseline and Week 12
  DLCO is a measurement of the ease of transfer for carbon monoxide molecules from alveolar gas to the hemoglobin of the red blood cells in the pulmonary circulation.
Change from baseline of patient reported outcomes by the University of California-San Diego (UCSD) Shortness of Breath Questionnaire (SOBQ) | Baseline and Week 12
  The UCSD SOBQ consists of 24 questions (21 assess severity of shortness of breath during specific activities of daily living; 3 additional items ask about limitations due to: shortness of breath, fear of harm from overexertion and fear of shortness of breath). Each question has a 6-point scale (0 = "not at all" to 5 = "maximal or unable to do because of breathlessness"), resulting in a total score ranging from 0 to 120 (a higher score represents a worse outcome).

OTHER OUTCOMES:
Change from baseline of FVC | Baseline and Week 6
Change from baseline of FVC | Baseline and Week 18
Change from baseline of DLCO | Baseline and Week 6
Change from baseline of DLCO | Baseline and Week 18
Change from baseline of patient reported outcomes by the UCSD SOBQ | Baseline and Week 6
Change from baseline of patient reported outcomes by the UCSD SOBQ | Baseline and Week 18

CONTACTS AND LOCATIONS:
Overall Officials: John Huetsch, M.D., Study Director — Endeavor Biomedicines
Locations (21):
- Australia (4):
  - Research Site, Liverpool, New South Wales
  - Research Site, Benowa, Queensland
  - Research Site, Box Hill, Victoria
  - Research Site, Clayton, Victoria
- Canada (2):
  - Research Site, Vancouver, British Columbia
  - Research Site, Sherbrooke, Quebec
- Malaysia (4):
  - Research Site, Batu Caves
  - Research Site, Kota Bharu
  - Research Site, Kuala Lumpur
  - Research Sire, Kuala Lumpur
- Mexico (6):
  - Research Site, Monterrey, Nuevo León
  - Research Site, San Nicolás de los Garza, Nuevo León
  - Research Site, Chihuahua City
  - Research Site, Mexico City
  - Research Site, Oaxaca City
  - Research Site, Puebla City
- South Korea (5):
  - Research Site (Namdong District), Incheon
  - Research Site (Bundang District), Seongnam
  - Research Site (Gangnam District), Seoul
  - Research Site (Seongbuk District), Seoul
  - Research Site (Songpa District), Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maher TM, Goldin JG, Hood J, Pitman J, de Los Rios M, Hobbs BP, Yu-Lin AB, Buendia-Roldan I, Thien F, Song JW, Perea PC, Ramirez-Rivera A, DiFrancesco A. Taladegib for the treatment of idiopathic pulmonary fibrosis (ENV-IPF-101): a multicentre, randomised, double-blind, placebo-controlled, phase 2a trial. Lancet Respir Med. 2025 Nov;13(11):1001-1010. doi: 10.1016/S2213-2600(25)00239-5. Epub 2025 Sep 30. PMID 41043447